CLINICAL TRIAL: NCT01643655
Title: Safety and Efficacy of Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Avascular Necrosis of the Femoral Head
Brief Title: Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Avascular Necrosis of the Femoral Head
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R-Bio (Industry)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSC-MSCs-AVN
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Avascular Necrosis of the Femoral Head
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Adipose Tissue Derived MSCs (Experimental)
  Interventions: Procedure: Autologous Adipose Tissue derived MSCs Transplantation

INTERVENTIONS:
Procedure: Autologous Adipose Tissue derived MSCs Transplantation — Into the Femoral Head infusion of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 1x10e8 cells/3mL

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with avascular necrosis of the femoral head.

ELIGIBILITY:
Inclusion Criteria:

* Age :18-70, males and females.
* Subjects who understand and sign the consent form for this study.
* Clinical diagnosis of nontraumatic avascular necrosis of the femoral head
* Steinberg stage I, II, ⅢA
* Patients whose lesion is more than 30% (by Kim's Method)

Exclusion Criteria:

* Patients who have collapsed femoral head
* Patient has had a Core Decompression or Multiple Drilling in the affected hip
* Patients who received osteoporosis medicines and parathyroid hormone drugs
* Taking medications that use the immunosuppressive drugs and cytotoxic agents or unable to discontinue their use for the duration of the study
* Taking medications that use the adrenocortical hormone drugs or unable to discontinue their use for the duration of the study
* Subject unable to undergo MRI (i.e. patients with pace-maker, metallic hip prosthetic implants)
* Women who are pregnant or breast feeding or planning to become pregnant during the study.
* Positive serology for HIV and hepatitis
* Serious pre-existing medical conditions like Cardiovascular Diseases, Cancer, Renal Diseases, Endocrine Diseases and Autoimmune Diseases
* Participation in another clinical trial or treatment with a different investigational product within 3 months prior to inclusion in the study.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging | 96 weeks
  To evaluate the change of treated femoral head using Magnetic Resonance Imaging (MRI) at 24 months post injection of MSCs.

SECONDARY OUTCOMES:
SPECT/CT | 96 weeks
  To evaluate the change of treated femoral head using SPEC/CT at 24 months post injection of MSCs.
Hip X-ray | 96 weeks
  To confirm the collapse of femoral head using Hip X-ray at 24 months post injection of MSCs.
HHS (Harris Hip Score) | 96 weeks
  To evaluate the change of treated femoral head using Harris Hip Score at 24 months post injection of MSCs.
WOMAC (Western Ontario and McMaster Universities) Index | 96 weeks
  To evaluate the change of treated femoral head using WOMAC Index at 24 months post injection of MSCs.
UCLA (University of California Los Angeles) hip questionnaire | 96 weeks
  To evaluate the change of treated femoral head using UCLA hip questionnaire at 24 months post injection of MSCs.
Safety evaluation | 96 weeks
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kang-Sup Yoon, M.D. & Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea